CLINICAL TRIAL: NCT04899882
Title: Physical Fitness Impact of Early Physiotherapy Intervention With a Standardized Exercise Therapy Program in Adult Patients Receiving Intensive Induction Chemotherapy for Treatment of Acute Leukemia During Extended Hospitalization. Randomized Controlled Superiority Trial in Parallel Arms, Multicentric (KinHémo)
Brief Title: Physical Fitness Impact of Early Physiotherapy Intervention With a Standardized Exercise Therapy Program in Adult Patients Receiving Intensive Induction Chemotherapy for Treatment of Acute Leukemia During Extended Hospitalization.
Acronym: KinHémo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49RC20_0030
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Acute Leukemia
Keywords: sarcopenia; exercise; cancer related fatigue
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- KinHémo group (Experimental)
  Interventions: Other: KinHémo

INTERVENTIONS:
Other: KinHémo — Evaluation and cardiovascular training, combination of resistance and flexibility training
  Arms: KinHémo group

SUMMARY:
This study aimed to investigate the impact of Physical therapy in adult patients receiving intensive induction chemotherapy for the treatment of acute leukemia during prolonged hospitalization. The study cohort included 150 patients. Primary objective is to compare the effect of a standardized rehabilitation program on physical deconditioning. This study has several secondary objectives of comparing and analyzing the status of sarcopenia, muscle strength, physical performance and the psychic dimension of this intervention. The 6 minutes walking test, Handgrip strength, impedance measurement, computed tomography, Short Physical Performance were used as measures of physical function. Hospital Anxiety and Depression Scale and European Organization for the Research and Treatment of Cancer-Quality of Life-Questionnaire-30 (EORTC-QLQ-30) were used as measures of depression and anxiety and quality of life of cancer patients. To investigate the impact of physical therapy, patients were assigned to the physical therapy group (experimental group) or the control group.These results will thus make it possible to promote access to physiotherapy and rehabilitation care, from diagnosis and during hospitalization, and to standardize practices.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient >18 years
* Patient with acute leukemia eligible to receive intensive chemotherapy (induction phase) with predictable deep bone marrow aplasia (polynuclear neutrophils <500mm3 for more than 8 days) requiring prolonged hospitalization with room confinement.
* Patient having signed the informed consent to participate in the study

Exclusion Criteria:

* Patient with disabilities or contraindications (significant cognitive or psychiatric disorders, significant cardiac or pulmonary pathology, neurological, joint, orthopedic or medical condition, etc.) following an exercise therapy program and carrying out follow-up defined by the protocol and in particular the physical performance tests.
* Active bleeding, acute thrombosis, ischemia, hemodynamic instability or uncontrolled pain
* No understanding of the French language
* Pregnant women, parturients and nursing mothers
* Persons deprived of their liberty by judicial or administrative decision
* People under duress psychiatric care
* Persons subject to legal protection
* Persons unable to express their consent
* Person not affiliated to a health insurance scheme or not beneficiary of a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2025-01-05 (Estimated); Study Completion 2025-03-05 (Estimated)

PRIMARY OUTCOMES:
The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity between V1 and V0 | The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity between V1 and V0
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.

SECONDARY OUTCOMES:
The physical performance assessed with Evolution of Short Physical Performance Battery | The worsening rate of sarcopenia defined either by the occurrence of a status of sarcopenia regardless of the stage or by moving from one sarcopenia stage's to another, 4 to 6 week after hospitalization
  Evolution of Short Physical Performance Battery measurements,
The muscle mass assessed with Bioelectrical impedance analysis | The worsening rate of sarcopenia defined either by the occurrence of a status of sarcopenia regardless of the stage or by moving from one sarcopenia stage's to another, 4 to 6 week after hospitalization
  Evolution of muscle mass by Bioelectrical impedance analysis
Anxiety and Depressive Disorders assessed with the Hospital Anxiety and Depression Scale | Hospital Anxiety and Depression Scale and European Organization for the Research
  Assessment of anxiety and depressive disorders
Evolution of activities of daily living assessed with Treatment of Cancer-Quality of Life Questionnaire-30 | The comparison visit 0 versus Visit 1 bis 10 to 15 days after discharge from hospital for induction
  Treatment of Cancer-Quality of Life Questionnaire-30 were used as measures of quality of life of cancer patients
muscle strength assessed with dynamometer and standing up test chair | The worsening rate of sarcopenia defined either by the occurrence of a status of sarcopenia regardless of the stage or by moving from one sarcopenia stage's to another, 4 to 6 week after hospitalization
  Evolution of muscle strength by measuring grip strength by dynamometer, evolution of the muscle strength of the lower limbs by standing up test chair
Rate of patients with at least one complication | The rate of patients with at least one complication is used as the outcome by wich to compare of effect of a standardized exercise therapy program versus practice current after 4-6 weeks hospitalization
  The comparison of the effect of a standardized exercise therapy program versus practice current hospitalization for the induction phase of chemotherapy: Complications of all types (pressure sore, infection, stay in intensive care).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Angers, Angers
  - CHU Brest, Brest
  - CHU Nantes, Nantes
  - CHU Tours, Tours